CLINICAL TRIAL: NCT00664066
Title: A Non-Interventional, Post-Authorisation Study to Assess Adverse Events and Drug Utilisation Among Chronic Kidney Disease Patients Treated With DYNEPO
Brief Title: DELFT (Dynepo Evaluation of Long-Term Follow-Up Treatment)
Acronym: DELFT
Status: Terminated | Type: Observational
Why Stopped: The termination of the study is not linked to a product recall or result of any safety signal. Rather it was sponsor's commercial decision to withdraw the MA
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SPD490-404
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Results first posted 2009-09-28 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-05

CONDITIONS: Anemia; Kidney Diseases; Renal Failure, Chronic; Kidney Failure, Chronic
MeSH Terms: conditions — Anemia; Kidney Diseases; Kidney Failure, Chronic | interventions — Erythropoietin; epoetin delta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: DYNEPO (epoetin delta) — dose, dose frequency, route of administration (iv or sc) and duration will be determined by the investigator according to their normal prescribing habits, as this is an observational study

SUMMARY:
This is a post-authorisation safety study to assess the incidence and severity of all pre-defined cardiovascular events in patients treated with DYNEPO, as well as to detect & describe less common adverse drug reactions, and to summarise DYNEPO drug utilisation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients must have established Chronic Kidney Disease (CKD) and be willing and able to provide written informed consent.
* Patients must already be receiving DYNEPO treatment at time of study entry.
* Patients who are likely to receive DYNEPO for at least 1 year.

Exclusion Criteria:

* Known intolerance to EPO of any of its excipients
* Known of suspected Pure Red Cell Aplasia (PRCA)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with established Chronic Kidney Disease
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2008-04-25 (Actual); Primary Completion 2008-07-30 (Actual); Study Completion 2008-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Germany (2):
  - Nephrologische Zentrum Villingen-Schwenningen, Villingen-Schwenningen, Baden-Wurttemberg
  - Hanse-Klinikum Stralsund, Stralsund

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated on July 31, 2008 as a result of a decision by Shire Pharmaceutical to permanently cease marketing Dynepo and withdraw the Marketing Authorisation. The decision was for commercial reasons, it was not the result of any safety signal.
Pre-assignment Details: The decision to enrol a subject was not to be made until after the decision on erythropoietin therapy had been made by the physician and drug had been prescribed. Physicians were to manage subjects according to their local practices and protocols.
Groups:
- Dynepo: Epoetin delta dose, dose frequency, route of administration (iv or sc) and duration will be determined by the investigator according to their normal prescribing habits
Period: Overall Study
Arm/Group | Dynepo
Started | 3
Completed | 0
Not Completed | 3
Not completed — Study terminated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Dynepo
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 57.0 (0.0) [57 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 3

OUTCOME MEASURES:

1. Primary Outcome: Assess the Incidence and Severity of All Predefined Cardiovascular Events in Subjects Treated With Dynepo
Description: This study was terminated on July 31, 2008 as a result of a decision by Shire Pharmaceutical to permanently cease marketing Dynepo and withdraw the Marketing Authorisation. The decision was for commercial reasons, it was not the result of any safety signal.
Time Frame: up to 3 years
Population: This study was terminated on July 31, 2008 as a result of a decision by Shire Pharmaceutical to permanently cease marketing Dynepo and withdraw the Marketing Authorisation. The decision was for commercial reasons, it was not the result of any safety signal.
Arm/Group | Dynepo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Dynepo
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
This study terminated early due to a decision by Shire Pharmaceuticals to permanently cease marketing Dynepo due to commercial reasons, it was not the result of any safety signal. Not enough subjects completed the study to do any efficacy analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.